CLINICAL TRIAL: NCT05276752
Title: Short- and Long-term Health Adverse Outcomes Associated With Nutrition Disorders and Nutrition Related Conditions in Hospitalized Older People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Head of geriatry department, Brugmann University Hospital
Other Study IDs: CHUB-Nutrition disorders
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition is associated with health adverse outcomes such as higher risk of mobility disability, falls and, fractures and higher mortality. Malnutrition had been defined as "a state resulting from lack of intake or uptake of nutrition that leads to altered body composition (decreased fat free mass) and body cell mass leading to diminished physical and mental function and impaired clinical outcome from disease". In 2018, the European Society for Clinical Nutrition and Metabolism (ESPEN) revisited nutrition and nutrition-related conditions definitions in the ESPEN guidelines on definitions and terminology of clinical nutrition based on the findings of the last decades. Nutrition disorders and nutrition related conditions were divided in 5 categories: Malnutrition/undernutrition, sarcopenia and frailty, overweight and obesity, micronutrients abnormalities, and refeeding syndrome. The definition of malnutrition based on the Global Leadership Initiative on Malnutrition (GLIM) criteria is globally accepted by de scientific community since this was launched in 2019. The presence of at least one phenotypic (i.e., nonintentional weight loss, low body mass index or low muscle mass) and one etiologic criterion (i.e., reduced food intake or inflammation) were required to define malnutrition.

Malnutrition is a common pathological condition in older adults that can further influence and aggravate health-related muscle decline. Sarcopenia is known as a natural progressive decline in skeletal muscles occurring with age, with an age-related decline in muscle strength. According to the criteria published in 2019 by the European Working Group on Sarcopenia in Older People (EWGSOP2), this process is defined by the presence of low muscle strength and low muscle mass.

Patients in acute care are likely to present higher stay and risk of mortality. However, the mortality have rarely been applied in acute care, due to difficulties to administer Dual X-ray Absorptiometry (DXA), the gold standard method for muscle mass in acute care. Pragmatic approaches to assess nutrition and nutrition-related condition are urgently needed to provide better quality of care in clinical practice in geriatric medicine.

The primary objective of this study is to determine the impact of nutrition disorders and nutrition-related conditions at baseline (admission in hospitalization) on the all-causes mortality risk in hospitalized older people.

Secondarily, this study evaluates their impact on other health adverse outcomes: falls, fractures, rehospitalization, institutionalization, all-cause admission in intensive care, length of hospital stay, length of ventilation and USI stay.

Finally, the diagnostic performance indicators of the Mini Nutritional Assessment (MNA-SF) and the Geriatric Nutritional Risk Index (GNRI) for malnutrition assessment following the GLIM criteria were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥60 and over admitted to the geriatric healthcare unit and/or the COVID-19 unit of the CHU Brugmann Hospital, between 01/01/2016 and 12/10/2021.
* Patients who had the assessment of nutrition disorders and/or nutrition related conditions available during their hospital admission.

Exclusion Criteria:

- No exclusion criteria based on demographical or medical data were applied.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥60 and over admitted to the geriatric healthcare unit and/or the COVID-19 unit of the CHU Brugmann Hospital, between 01/01/2016 and 12/10/2021.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | From 2016 till 2021
  Vital status (death/alive)

SECONDARY OUTCOMES:
Falls | From 2016 till 2021
  Falls (yes/no)
Fractures of upper and lower limbs and/or hip and/or vertebrae | From 2016 till 2021
  Fractures of upper and lower limbs and/or hip and/or vertebrae (yes/no)
Re-hospitalization | From 2016 till 2021
  Unplanned readmission in hospital (yes/no)
Institutionalization | From 2016 till 2021
  Institutionalization (yes/no)
All-cause admission in intensive care | From 2016 till 2021
  All-cause admission in intensive care (yes/no)
Mechanical ventilation | From 2016 till 2021
  Mechanical ventilation (yes/no)
Length of hospital stay time from admission to discharge | From 2016 till 2021
  Length of hospital stay time from admission to discharge
Sensitivity | From 2016 till 2021
  Diagnostic performance indicators: the ability of a screening test to identify malnourished patients according to the GLIM criteria.
Specificity | From 2016 till 2021
  Diagnostic performance indicators: the ability of a screening test to identify non-malnourished patients according to the GLIM criteria.
Positive predictive value (PPV) | From 2016 till 2021
  Positive predictive value is the proportion of positive screening test results that are true positives for the diagnosis of malnutrition according to GLIM criteria.
Negative predictive value (NPV) | From 2016 till 2021
  Negative predictive value (NPV) is the proportion of negative screening test results that are true negative for the diagnosis of malnutrition according to the GLIM criteria.
Area under the ROC curve (AUC) | From 2016 till 2021
  A measure of the precision of a quantitative diagnostic test, which gives equal weight to sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Claessens, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Meester D, Goossens M, Marco E, Claessens M, Gautier J, Annweiler C, Lieten S, Benoit F, Surquin M, Sanchez-Rodriguez D. Evaluation of the Geriatric Nutritional Risk Index in predicting mortality in older patients with COVID-19 in the AgeBru cohort. Clin Nutr ESPEN. 2023 Oct;57:65-72. doi: 10.1016/j.clnesp.2023.06.025. Epub 2023 Jun 25. PMID 37739719